CLINICAL TRIAL: NCT04819308
Title: Substrate Utilization in Pre-pubertal Children During Submaximal Exercise and Rest ("SUPER Kids")
Brief Title: Differences in Nutrient Use During Exercise Between Children of Varying Body Mass Indices and Fitness Levels
Acronym: SUPERkids
Status: Active, not recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 261146
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-09

CONDITIONS: Obesity
Keywords: Children; Kids; Physical Activity; Exercise; Substrate Oxidation; Fat Oxidation; Carbohydrate Oxidation; Fitness; Nutrient; Obesity
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children who have previously participated in the study "MI Energy" will be invited to participate in "SUPER kids". Investigators want to better understand differences in nutrient use (e.g., fatty acid and carbohydrate) during rest and exercise in children of varying body types and activity levels.

DETAILED DESCRIPTION:
We will examine fatty acid oxidation (FAO) and carbohydrate (CHO) oxidation at rest and during exercise in children of all body types and activity levels.

Children 8-11 years old who have done the "MI Energy" study will participate. Up to 80 children will be recruited to participate in this study at Arkansas Children's Nutrition Center (ACNC).

They will be asked to attend three study visits (baseline, and two exercise visits). For the exercise visits, they will follow a diet plan and be encouraged to avoid certain foods and activities.

Children will do two testing days with the following measures:

* Urine (pee) will be collected
* Body weight and height
* Exercise test on the bike - children will ride a stationary bike at a set intensity and at an intensity relative to their previous bike test during the study "MI Energy". The order in which they bike will be random. Before and during biking, children will wear a mask that will measure the gases in their breath and a monitor that will measure heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Boys or girls
* Ages 8-11 years
* All races
* All ethnicities
* All BMIs
* Children who completed a dual-energy x-ray absorptiometry (DXA) scan during "MI Energy" (IRB Protocol: 260376)
* Children who completed a fitness test during "MI Energy" (IRB Protocol: 260376) and achieved peak oxygen uptake (VO2 peak)
* All fitness levels [VO2 peak already determined under "MI Energy" (IRB Protocol: 260376)]
* Children whose parents consented to the following in the "MI Energy" (IRB Protocol: 260376) study:

A) be contacted about future follow-up studies to "MI Energy", and having the data that is collected about their child in "MI Energy" being used also in these follow-up studies; and B) information collected in the "MI Energy" study may be used in future research related to bioenergetics (for example, blood cell mitochondria function), nutrition, obesity, cardiovascular health, or development; and C) any biological samples collected in the "MI Energy" study may be used in future research related to bioenergetics (for example, blood cell mitochondria function), nutrition, obesity, cardiovascular health, or development.

Exclusion Criteria:

* Participants who have been excluded from participation in the study "MI Energy" (IRB Protocol: 260376).
* Participants whose parents report any change in medical history that may potentially affect participation and/or study outcomes as determined by PI.
* Participants whose parents report food allergies or intolerances to nuts, wheat, dairy, or eggs.
* Participants whose parents report unwillingness to follow dietary standardization.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children ages 8-11, who have previously participated in the study "MI Energy".
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Substrate Oxidation | 24 months
  Carbohydrate oxidation and fatty acid oxidation quantified using breath samples measured by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Borsheim, PhD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

REFERENCES:
- See also: Arkansas Children's Nutrition Center webpage — https://medicine.uams.edu/pediatrics/research/acnc/

DOCUMENTS (1):
  • Informed Consent Form (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT04819308/ICF_000.pdf